CLINICAL TRIAL: NCT03385980
Title: Donation of Post Mortem Tumor Tissues to Unravel Cancer Heterogeneity
Brief Title: Donation of Post Mortem Tumor Tissues
Acronym: DONUM
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Collaborators: University of Turin, Italy (Other); Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 90/317/16
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: NSCLC Stage IV; CRC; CUP
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary and metastatic tissues and peripheal blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-mortem patients: Post-mortem oncological patients (within 2-6 hrs from death, maximum time for tissue preservation).
  Interventions: Other: Proteomic analysis

INTERVENTIONS:
Other: Proteomic analysis — Proteomic analysis of tissues collected from all sites of disease, guided by either imaging performed prior to the patient's death or post-mortem findings. Peripheral blood mononuclear cells (PBMC) will be collected with the purpose of identifying somatic changes occurring specifically in the tumor cells and not in normal DNA of the same patient.

SUMMARY:
DONUM is an observational prospective independent protocol for patients with advanced lung cancer, colorectal cancer or cancer of unknown primary, willing to donate their tumor tissue samples post mortem for biomedical research purposes. All patients who fulfill the inclusion criteria will be eligible for the study after giving their Informed consent. Informed Consent will be obtained in two steps. During the pre-information step patients will be acquainted with the existence of a post-mortem cancer tissue donation research program governed by the DONUM protocol. If the patients manifest interest to participate into the program (in writing) during the pre-information step, they will proceed to step 2 and undergo the final informed consent process.

DETAILED DESCRIPTION:
Despite the recent technological advancement in genomic and proteomic, the molecular understanding of clonal evolution in solid tumor patients is hampered by intra tumor heterogeneity (ITH), while remaining essential to the effective treatment of patients. Recent evidence suggests that branched evolutionary tumor growth may contribute to ITH both within a primary tumor and between primary and metastatic tumors. To study the full extent and consequences of ITH, and grasp clonal evolution, the investigators need to have access not only to circulating biomarkers (circulating tumor DNA) but also, simultaneously and separately, to the primary tumor and all its derived metastases. However multiple biopsies in live patients are neither medically feasible, nor ethical acceptable. A lesser known tissue collection method is through rapid tissue donation (RTD), which is the procurement of 'fresh' tissue within 2 hrs following the death of a patient. RTD-based research provides an effective way to investigate advance tumors biology in a manner not possible by any other means. With an RTD approach, the full extent and consequences of tumor heterogeneity can be evaluated by deep sequencing and global analysis of genetic alterations at the protein level of simultaneous core biopsies from several areas of the primary tumor and metastases and correlation with clinical outcome. To investigators' knowledge, no such studies have been done in Italy and are currently being pursued only in selected USA and UK cancer centers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed metastatic non-small cell lung cancer (NSCLC), colorectal cancer (CRC), CUP (cancer of unknown origin syndrome) with life expectancy less than or equal to 3/4 months;
* Age ≥18;
* Signed informed consent from patient to enter the study and to undergo post-mortem tissue sampling.

Exclusion Criteria:

* Medical, or psychological conditions that would preclude informed consent;
* History of high-risk infections (e.g. HIV-positive, hepatitis C, tuberculosis and Creutzfeldt-Jacob disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with confirmed metastatic non-small cell lung cancer (NSCLC), colorectal cancer (CRC), CUP (cancer of unknown origin syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Intratumor heterogeneity | within 2-6 hours post-mortem
  Procure primary and metastatic tissue of selected solid tumor patients shortly after death in order to investigate ITH (intratumor heterogeneity), using integrated genomic and proteomic analysis

SECONDARY OUTCOMES:
Potential impact on subsequent lines of therapy | within 2-6 hours post-mortem
  Study ITH as a results of anticancer drugs exposure in order to forecast its potential impact on subsequent lines of therapy
Circulating free tumor DNA | within 2-6 hours post-mortem
  Study how the genomic landscape provided by the determination of the circulating free tumor DNA (ctDNA) compare to the genomic landscape from all tumor tissues, considered as gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Siena, MD, Principal Investigator — Niguarda Cancer Center
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siravegna G, Lazzari L, Crisafulli G, Sartore-Bianchi A, Mussolin B, Cassingena A, Martino C, Lanman RB, Nagy RJ, Fairclough S, Rospo G, Corti G, Bartolini A, Arcella P, Montone M, Lodi F, Lorenzato A, Vanzati A, Valtorta E, Cappello G, Bertotti A, Lonardi S, Zagonel V, Leone F, Russo M, Balsamo A, Truini M, Di Nicolantonio F, Amatu A, Bonazzina E, Ghezzi S, Regge D, Vanzulli A, Trusolino L, Siena S, Marsoni S, Bardelli A. Radiologic and Genomic Evolution of Individual Metastases during HER2 Blockade in Colorectal Cancer. Cancer Cell. 2018 Jul 9;34(1):148-162.e7. doi: 10.1016/j.ccell.2018.06.004. PMID 29990497